CLINICAL TRIAL: NCT03757637
Title: Yeur-Hur Lai, PhD, RN, School of Nursing, College of Medicine, National Taiwan University
Brief Title: Compare the Effects of NLSCP and Interactive ICT Supported HAP on Differentiate Diagnosed Thyroid Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 201712196RIND
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Differentiated Thyroid Cancer
Keywords: Thyroid cancer; Survivorship Care; Mobile applications; Mobile phone
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: There are various models of SCP, in general, the primary care physician model or nurse-led model are generally being recognized for effective detecting patients' distress and recurrences, effective coordination and communication, and taking SCP as standard cancer care. In Taiwan, we take a large number of advanced DTC patients, it is important to integrate the SCP but also need to concern about the limited time in busy OPD clinics and patients' differences because of various physical or psychological conditions and needs. We will build up the contents and operable programs for two interventions groups: NLSCP and ICT supported HAP.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: This study was not fully blinded; however, the group allocation was concealed from the patient and primary researcher until after baseline assessments were completed. A primary researcher obtained patient consent, collected selfreported assessments, and if the patients were randomized to intervention group, the intervention trainer explained the exercise program to participants. The study statistician and data managers remained blinded at all times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General module (No Intervention): Control group will be "case manager care only" group. Eligible patients will also invite and receive their first time assessment as baseline during hospitalization. The usual cancer care group will receive routine cancer care in the inpatient wards through OPD visits.
- NLSCP (Experimental): NLSCP group will receive 5 section of NLSCP. Contents of scheduled intervention will be developed baed on the literature mentioned above. Ex 1 group, patients will receive at least 3 times face-to-face NLSCP, and two times by telephone calls for following up.
  Interventions: Other: NLSCP
- ICT supported HAP (Experimental): The ICT supported HAP group will receive information or counseling through mobile phone App as the schedule intervention time. For this group, patients will receive two face to face interventions in the first two sections (pre-discharge from hospital and 5th week post-op). It will be delivered by research nurse to intervene patients and help them to build up the App system. Research nurse will also help patients to be familiar with the operation system. The rest parts of the intervention will all through Apps in the scheduled time. Patients can raise their questions and concerns through APPs. Patients in the HAP can raise their concerns or questions through APP and receive interventions or answers through App interactively.
  Interventions: Other: ICT supported HAP

INTERVENTIONS:
Other: NLSCP — Phase II is a 6-month three-group randomized controlled trial with 12 month follow-up of its effects. In addition to receive hospital routine case manager care, patients in this groups will further receive either NLSCP (Exp-1). Patients will be provided the same major education and counseling contents for the first two section of interventions through face-by-face by trained research nurses at time of (1) first intervention: one day before hospital discharge in post-operation, and (2) second intervention: first OPD visit (first week after hospital discharge). This group will receive a face-to-face education or counseling by trained research nurse.
  Arms: NLSCP
Other: ICT supported HAP — Phase II is a 6-month three-group randomized controlled trial with 12 month follow-up of its effects. In addition to receive hospital routine case manager care, patients in the groups will further receive ICT supported HAP (Exp-2) intervention. For this groups, patients will be provided the same major education and counseling contents for the first two section of interventions through face-by-face by trained research nurses at time of (1) first intervention: one day before hospital discharge in post-operation, and (2) second intervention: first OPD visit (first week after hospital discharge). The group will receive the interactive mobile phone App.
  Arms: ICT supported HAP

SUMMARY:
Background: Despite the good prognosis of patients with differentiated thyroid carcinomas (DTC), the diagnosis of cancer, fear of cancer recurrence and its side effects might still bring impacts on patients' quality of life and daily function.

Purposes: This is a two-phase study. Phase I will aim to examine the current concerns of patients' physical-, psychological, care needs, and physical and psychological function in DTC patients within one year of diagnosis, and identify factors related to patients' physical and psychological functions. Phase II will be a three-group randomized control trail (RCT). The aims will be develop two intervention programs: Nurse-led Survivorship Care Program (NLSCP, Exp-1) and Information & Communication Technology (ICT) Supported Healthy Active Program (ICT supported HAP, Exp-2), and compare the effects of the two intervention groups and control group of their effects on the variables in the above mentioned four dimensions (physical, psychological, care needs, function) in newly diagnosed DTC patients receiving total thyroidectomy.

Methods: Phase I is a cross-sectional survey study and to examine the current status of physical distress (e.g., fatigue, pain), psychological distress (e.g., depression, body-image), care needs, and psychological & physical functions. Phase II is a 6-month three-group RCT with 12 month follow-up of its effects. There will have 5 intervention sections during the first 6 month. Control group will be case manager care only. The NLSCP will receive face-to-face or telephone education by trained nurse. The ICT supported HAP group will receive information or counseling through mobile phone App as the schedule intervention time. For both Exp groups, the first 2 sections of interventions will be all delivered face-to-face for helping them to be familiar with the operation system. Patients in the ICT supported HAP group can raise their concerns or questions through APP and receive intervention through App interactively. The outcomes will be assessed at 5 time points: time before first intervention (baseline assessment), 4-5 week before intervention, 3-, 6-, and 12 months.

Expected Outcome: We expect this study can help us better understanding DTC patients' impacts and care needs. The comparison of three groups of intervention will also help us to identify the best model to decrease distress and enhance life function for them.

DETAILED DESCRIPTION:
Phase I is a cross-sectional survey study (first year) with the specific aims to examine the current status of physical distress (fatigue, sleep dysfunction, other symptoms), psychological distress (fear of cancer recurrence, depression, body-image), care needs, and psychological & physical functions in DTC patients diagnosed within three years. We will also examine these factors of their relationship with physical and psychological function by short-form -12.

Phase II is a 6-month three-group randomized controlled trial with 12 month follow-up of its effects. Eligible subjects will be those newly diagnosed DTC patients with total thyroidectomy. A stratified randomization by age (age 45 as cut-off point) and gender would be conducted. Although the different intervention designs in the two intervention groups (NLSCP & ICT supported HAP). The three groups, control and two intervention groups (Exp-1 & Exp-2) will all receive the hospital routine and case manager's care. The three groups will receive baseline assessment before first intervention during hospitalization. We will first build up the contents and operable programs for two interventions groups: nurse-led survivorship care program (NLSCP/ Exp-1) and ICT supported HAP (ICT supported HAP/ Exp-2). Both intervention groups will also receive routine case manager care too. For both intervention groups, there will have 5 intervention sections during the first 6 month, including one day before hospital discharge post-operation, 5-6th week and 2-, 3-, 5- month post operation, known as intervention 1-5, respectively.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed DTC patients
* after received thyroid tumor excision operation (total thyroidectomy)

Exclusion Criteria:

* primary unknown
* conscious unclear
* recurrence or with bone meta

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety & Depression Scale (HADS) | For all groups, we will assess patients' outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital).
  The severity of lung cancer patients' anxiety and depression will be measured by the self-reporting HADS. The 14 items of HADS consists of two subscales, include 7 items anxiety and 7 items depression. The score of all items ranges from 0 (not at all) to 3 (always) and the total score of each subscale arerange from 0 to 21, a higher score indicates a higher level of anxiety or depression. Satisfactory psychometrics of the HADS has been shown in cancer populations in Taiwan (Chen et al. 2000).
Fear of Recurrence Inventory | For all groups, we will assess patients' outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital).
  The FoR-C is a Chinese version of the original FoR questionnaire. The FoR questionnaire consists of six statements with a five-point response scale from not at all (1), a little, sometimes (2), a lot , and all the time) and one statement with a response scale from 0 (not at all) to 10 (a great deal). The summary of FoR was range from 6 to 40. Higher score indicates a higher level of fear of recurrence. The significance of the FoR was indicated by patients' responses 'a lot' or 'all the time' for the first six statements and the score of 7-10 for the last item, in which case. Current study will use the same approach to determine the cut-off point of the FoR.
Body Image Scale (BIS) | For all groups, we will assess patients' outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital).
  The Body Image Scale (BIS) was developed to assess body image. The 10-item BIS comprised three subscales: affective (e.g. feeling feminine/masculine, physically attractive, or sexually attractive), behavioral (e.g. find it hard to look at youeself naked, avoid people because of appearance), and cognitive (e.g. satisfied with appearance, or with scar). Five items were presented positively and the others were presented negatively. Each item was scored from 0 (not at all) to 3 (very much). The higher overall summary score indicated more symptoms and distress. (Hopwood, Fletcher, Lee, & Al Ghazal, 2001) The BIS has been translated to Chinese and validated to be reliable in cancer patients in Taiwan. Cronbach's α was 0.84-0.94. (Chen, Liao, Chen, Chan, & Chen, 2012; Chen et al., 2017; Hung et al., 2017).
Fatigue Severity Inventory | For all groups, we will assess patients' outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital).
  The Fatigue Symptom Inventory (FSI) was developed to assess fatigue in patients with cancer. It's a 14-item self-reported measure designed to assess the intensity (four items), duration (two items), daily pattern (one item) and inference (seven items) of fatigue. The Items assessing intensity and interference are scored on an 11-point Likert-type scale (0 = not at all fatigued/ no inference at all; 10 = as fatigued as I could be/ extreme inference). Two items assessing duration are based on the number of days in the past week patients felt fatigue (0 - 7 days) and the percent of time each day fatigue was present (0 = none of the day; 10 = the entire day). (Hann, Denniston, & Baker, 2000; Hann et al., 1998) The Chinese version of FSI has been validated in patients with cancer and its Cronbach's α was 0.92. (Chou, Lai, Wang, & Shun, 2017; Shun, Beck, Pett, & Berry, 2006; Shun, Beck, Pett, & Richardson, 2007).
Pittsburgh's Sleep Index | For all groups, we will assess patients' outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital).
  The PSQI was developed by Buysee in 1989, is used to assess sleep quality on participants' sleep experiences during the past week (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989). Iincluding seven component scores which are sleep duration, sleep disturbances, sleep latency, daytime functioning, habitual sleep efficiency, sleep quality, and sleep medication. The total PSQI score range is from 0 to 21, and the higher the worse of the sleep. If the total PSQI score is more than 5, the result means the person has sleep problems (Buysse et al., 1989; He et al., 2015; Van Onselen et al., 2010). In Chinese-PSQI, Cronbach's a coefficient for the hospital sample and test-retest reliability were 0.83 and 0.85, respectively (Tsai et al., 2005). Normal and problem sleepers (PSQI total score≦5 or >5) had 90% of sensitivity and 87% of specificity in original questionnaire (Buysse et al., 1989) and had 98% of sensitivity and 55% of specificity in Chinese version questionnaire (Tsai et al., 2005).
Brief Supportive Care Needs Survey (SCNS-9) | For all groups, we will assess patients' outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital).
  The unmet needs of lung cancer patient will be measured by 9 items SCNS. It consists of 5 domains, include psychological, health system and information, daily living, patient care and sexuality domain. Response options "No need, not applicable (1); No need, satisfied (2); Low need (3); Moderate need (4); High need (5). The sum of item scores within each domain will be calculated and the scores will be transformed to a standardized score 0 to 100, higher score indicate more unmet needs (Girgis, Stojanovski, Boyes, King, & Lecathelinais, 2011). The higher scores representing more unmet needs (McElduff, Boyes, Zucca, & Girgis, 2004). A previous study reported the construct reliability and construct validity of this instrument (Girgis et al, 2011). The Chinese SCNS34 has acceptable psychometric properties in previous lung cancer studies (Liao et al., 2011; Shun et al., 2014).
Short Form 12 (SF-12) | For all groups, we will assess patients' outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital).
  The Short Form-12 (SF-12) Health Survey is a shortened version of the 36-item Short Form Health Survey with 12 items. It's a generic and validated self-reported health-related quality-of-life questionnaire. The SF-12 consists of eight-scale scores and two summary measures: physical and mental component summary measures (PCS and MCS). It includes two items on physical functioning, two items on role physical, one item on bodily pain, one item on general health, one item on vitality, one item on social functioning, two items on role emotional, and two items on mental health. (Busija et al., 2011; Fong et al., 2010; Ware et al., 1996) The SF-12 scores are calculated by summing the raw scores and transform to a 0-100 scale. The higher score indicated better health. (Busija et al., 2011) The previous study reported Cronbach's α for the Chinese version of the PCS was 0.62-0.83 and the MCS was 0.75-0.76. (Chou, Lai, Wang, & Shun, 2017; Fong et al., 2010).
Symptom Severity Scale (SSS) | For all groups, we will assess patients' outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital).
  Symptom Severity Scale was developed to assess patients' symptom severity, and it will be modified to assess disease and treatment-related symptoms in DTC patients. Each item of this 23-item SSS is rated from 0 to 10, with 0 indicating "no such symptom at all" and 10 indicating "extreme severity of the symptom." The SSS has been validated as a reliable scale (Chen et al., 2010; Chen et al., 2013).
Impact of Event Scale-Revised (IES-R) | For all groups, we will assess patients' outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital).
  The IES is developed by Horowitz et al. (1979) and it was further revised. The IES-R can directly assess the impact of cancer to patients and it is based on mechanisms of people's dealing with calamitous life events. This instrument includes two psychological dimensions: intrusion and avoidance, and it has good psychometrics characteristics. The IES is scored on a 0-5 scale with the higher the score, the more the intrusion and the greater the avoidant tendency or avoidance (Sundin & Horowitz, 2003).
Illness Perception Questionnaire (IPQ-M) | For all groups, we will assess patients' outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital).
  The Illness Perception Questionnaire (IPQ) was developed by Broadbent, Petrie, Main and Weinman (2006) and it is for measuring patients' perception about their illness. Also the IPQ has been proven a good psychometric measurement. The IPQ was later modified by Grunfeld, and Cooper (2010) to assess cancer patients' concerns, perception and barriers of their return to work. The 26-item IPQ-M which consists of two major dimensions: (1) the impacts of cancer and its treatment on work, and (2) illness perceptions in relation to work was an 8-point Likert's scale scoring from 0 to 7 with the higher score indicating more concerns or barriers about RTW.

CONTACTS AND LOCATIONS:
Overall Officials: Yeur-Hur Lai, Professor, Study Chair — School of Nursing, College of Medicine, National Taiwan University
Locations (1):
- Department of Surgery, National Taiwan University Hospital, No.7, Chung-Shan South Road, Taipei, TAIWAN, R.O.C., Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen ML, Chang HK, Yeh CH. Anxiety and depression in Taiwanese cancer patients with and without pain. J Adv Nurs. 2000 Oct;32(4):944-51. PMID 11095234
- [Background] Hopwood P, Fletcher I, Lee A, Al Ghazal S. A body image scale for use with cancer patients. Eur J Cancer. 2001 Jan;37(2):189-97. doi: 10.1016/s0959-8049(00)00353-1. PMID 11166145
- [Background] Chen CL, Liao MN, Chen SC, Chan PL, Chen SC. Body image and its predictors in breast cancer patients receiving surgery. Cancer Nurs. 2012 Sep-Oct;35(5):E10-6. doi: 10.1097/NCC.0b013e3182336f8b. PMID 22067694
- [Background] Chen SC, Huang BS, Lin CY, Fan KH, Chang JT, Wu SC, Lai YH. Psychosocial effects of a skin camouflage program in female survivors with head and neck cancer: A randomized controlled trial. Psychooncology. 2017 Sep;26(9):1376-1383. doi: 10.1002/pon.4308. Epub 2016 Dec 2. PMID 27859893
- [Background] Hung TM, Lin CR, Chi YC, Lin CY, Chen EY, Kang CJ, Huang SF, Juang YY, Huang CY, Chang JT. Body image in head and neck cancer patients treated with radiotherapy: the impact of surgical procedures. Health Qual Life Outcomes. 2017 Aug 23;15(1):165. doi: 10.1186/s12955-017-0740-7. PMID 28830456
- [Background] Hann DM, Denniston MM, Baker F. Measurement of fatigue in cancer patients: further validation of the Fatigue Symptom Inventory. Qual Life Res. 2000;9(7):847-54. doi: 10.1023/a:1008900413113. PMID 11297027
- [Background] Hann DM, Jacobsen PB, Azzarello LM, Martin SC, Curran SL, Fields KK, Greenberg H, Lyman G. Measurement of fatigue in cancer patients: development and validation of the Fatigue Symptom Inventory. Qual Life Res. 1998 May;7(4):301-10. doi: 10.1023/a:1024929829627. PMID 9610214
- [Background] Chou YY, Lai YH, Wang SS, Shun SC. Impact of Fatigue Characteristics on Quality of Life in Patients After Heart Transplantation. J Cardiovasc Nurs. 2017 Nov/Dec;32(6):551-559. doi: 10.1097/JCN.0000000000000400. PMID 28306705
- [Background] Shun SC, Beck SL, Pett MA, Berry PH. Psychometric testing of three Chinese fatigue instruments in Taiwan. J Pain Symptom Manage. 2006 Aug;32(2):155-67. doi: 10.1016/j.jpainsymman.2006.02.011. PMID 16877183
- [Background] Shun SC, Beck SL, Pett MA, Richardson SJ. Assessing responsiveness of cancer-related fatigue instruments: distribution-based and individual anchor-based methods. Oncologist. 2007 Apr;12(4):495-504. doi: 10.1634/theoncologist.12-4-495. PMID 17470692
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] He Y, Meng Z, Jia Q, Hu F, He X, Tan J, Zhang G, Li X, Zhang J, Zhang Q, Liu L, Zhao L, Li J, Wang Y, Qian Y, Hou S, Liu H, Wang S, Wang R, Zheng W, Hu T, Liu N, Upadhyaya A, Liu Y. Sleep Quality of Patients with Differentiated Thyroid Cancer. PLoS One. 2015 Jun 17;10(6):e0130634. doi: 10.1371/journal.pone.0130634. eCollection 2015. PMID 26083787
- [Background] Van Onselen C, Dunn LB, Lee K, Dodd M, Koetters T, West C, Paul SM, Aouizerat BE, Wara W, Swift P, Miaskowski C. Relationship between mood disturbance and sleep quality in oncology outpatients at the initiation of radiation therapy. Eur J Oncol Nurs. 2010 Dec;14(5):373-9. doi: 10.1016/j.ejon.2009.12.002. Epub 2010 Jan 18. PMID 20080444
- [Background] Tsai PS, Wang SY, Wang MY, Su CT, Yang TT, Huang CJ, Fang SC. Psychometric evaluation of the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI) in primary insomnia and control subjects. Qual Life Res. 2005 Oct;14(8):1943-52. doi: 10.1007/s11136-005-4346-x. PMID 16155782
- [Background] Girgis A, Stojanovski E, Boyes A, King M, Lecathelinais C. The next generation of the supportive care needs survey: a brief screening tool for administration in the clinical oncology setting. Psychooncology. 2012 Aug;21(8):827-35. doi: 10.1002/pon.1973. Epub 2011 Apr 12. PMID 21484938
- [Background] Liao YC, Liao WY, Shun SC, Yu CJ, Yang PC, Lai YH. Symptoms, psychological distress, and supportive care needs in lung cancer patients. Support Care Cancer. 2011 Nov;19(11):1743-51. doi: 10.1007/s00520-010-1014-7. Epub 2010 Oct 15. PMID 20949362
- [Background] Shun SC, Yeh KH, Liang JT, Huang J, Chen SC, Lin BR, Lee PH, Lai YH. Unmet supportive care needs of patients with colorectal cancer: significant differences by type D personality. Oncol Nurs Forum. 2014 Jan 1;41(1):E3-11. doi: 10.1188/14.ONF.E3-E11. PMID 24368251
- [Background] Busija L, Pausenberger E, Haines TP, Haymes S, Buchbinder R, Osborne RH. Adult measures of general health and health-related quality of life: Medical Outcomes Study Short Form 36-Item (SF-36) and Short Form 12-Item (SF-12) Health Surveys, Nottingham Health Profile (NHP), Sickness Impact Profile (SIP), Medical Outcomes Study Short Form 6D (SF-6D), Health Utilities Index Mark 3 (HUI3), Quality of Well-Being Scale (QWB), and Assessment of Quality of Life (AQoL). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S383-412. doi: 10.1002/acr.20541. No abstract available. PMID 22588759
- [Background] Fong DY, Lam CL, Mak KK, Lo WS, Lai YK, Ho SY, Lam TH. The Short Form-12 Health Survey was a valid instrument in Chinese adolescents. J Clin Epidemiol. 2010 Sep;63(9):1020-9. doi: 10.1016/j.jclinepi.2009.11.011. Epub 2010 Mar 1. PMID 20189764
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Chen SC, Lai YH, Liao CT, Lin CC, Chang JT. Changes of symptoms and depression in oral cavity cancer patients receiving radiation therapy. Oral Oncol. 2010 Jul;46(7):509-13. doi: 10.1016/j.oraloncology.2010.02.024. Epub 2010 Mar 21. PMID 20308004
- [Background] Chen SC, Lai YH, Liao CT, Chang JT, Lin CY, Fan KH, Huang BS. Supportive care needs in newly diagnosed oral cavity cancer patients receiving radiation therapy. Psychooncology. 2013 Jun;22(6):1220-8. doi: 10.1002/pon.3126. Epub 2012 Jun 25. PMID 22730021
- [Background] Zilberg NJ, Weiss DS, Horowitz MJ. Impact of Event Scale: a cross-validation study and some empirical evidence supporting a conceptual model of stress response syndromes. J Consult Clin Psychol. 1982 Jun;50(3):407-14. doi: 10.1037//0022-006x.50.3.407. No abstract available. PMID 7096742
- [Background] Horowitz M, Wilner N, Alvarez W. Impact of Event Scale: a measure of subjective stress. Psychosom Med. 1979 May;41(3):209-18. doi: 10.1097/00006842-197905000-00004. PMID 472086
- [Background] Sundin EC, Horowitz MJ. Horowitz's Impact of Event Scale evaluation of 20 years of use. Psychosom Med. 2003 Sep-Oct;65(5):870-6. doi: 10.1097/01.psy.0000084835.46074.f0. PMID 14508034
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Grunfeld EA, Low E, Cooper AF. Cancer survivors' and employers' perceptions of working following cancer treatment. Occup Med (Lond). 2010 Dec;60(8):611-7. doi: 10.1093/occmed/kqq143. Epub 2010 Sep 20. PMID 20855546